CLINICAL TRIAL: NCT00605683
Title: A Phase III, Double-blind, Placebo-controlled Randomised Trial to Determine the Efficacy and Safety of a Low (50 mg/Day) and High (100 mg/Day) Dose of Safinamide, as add-on Therapy, in Subjects With Early Idiopathic Parkinson's Disease Treated With a Stable Dose of a Single Dopamine Agonist
Brief Title: MOTION, Safinamide in Early IPD, as add-on to Dopamine Agonist
Acronym: MOTION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27918; 63,901; EudraCT: 2007-002963-28
Record Dates: First submitted 2007-12-19; First posted 2008-01-31 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-03

CONDITIONS: Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide; Apomorphine; Bromocriptine; Pramipexole; ropinirole; Cabergoline; Lisuride; Pergolide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Active Comparator): 50 mg/day Safinamide
  Interventions: Drug: Safinamide (as add-on therapy)
- 2 (Active Comparator): Safinamide 100mg/day
  Interventions: Drug: Safinamide (as add-on therapy)
- 3 (Placebo Comparator): Placebo 0mg/Safinamide
  Interventions: Drug: Safinamide (as add-on therapy)

INTERVENTIONS:
Drug: Safinamide (as add-on therapy) — Safinamide, (S)-(+)-2-[4-(3-fluorobenzyloxy) benzylamino] propanamide methanesulfonate, is an a-aminoamide derivative
  Other Names: Apokyn; Parlodel; Mirapex; Requip; Cabergoline (not approved in US); Lisuride (not approved in US); Pergolide (withdrawn from US Market March 2007)
  Arms: 1
Drug: Safinamide (as add-on therapy) — Safinamide add-on therapy with subjects with IPD treated with single dopamine agonist
  Other Names: Apokyn; Parlodel; Mirapex; Requip; Cabergoline (not approved in US); Lisuride (not approved in US); Pergolide (withdrawn from US Market March 2007)
  Arms: 2
Drug: Safinamide (as add-on therapy) — Safinamide add-on therapy with subjects with IPD treated with single dopamine agonist
  Other Names: Apokyn; Parlodel; Mirapex; Requip; Cabergoline (not approved in US); Lisuride (not approved in US); Pergolide (withdrawn from US Market March 2007)
  Arms: 3

SUMMARY:
Parkinson's disease is a major neurodegenerative disorder in which there is a progressive loss of nigrostriatal dopaminergic neurons. The understanding that PD is a syndrome of dopamine (DA) deficiency led to the introduction in the clinical practice of L-dopa, a precursor of DA that crosses the blood brain barrier, and also to the use of selective inhibitors of MAO B, the major DA metabolising enzyme in man.

This is a double-blind, placebo-controlled, parallel-group, randomised, multi-centre, multi national, Phase III trial, comparing two doses of safinamide (50 and 100 mg p.o. q.a.m.) versus placebo as add-on therapy to a stable dose of a single dopamine agonist in subjects with early idiopathic Parkinson's Disease.

The principal efficacy measure, i.e., change in mean value of UPDRS - Section III total score from baseline to endpoint, was chosen based on regulatory guidance and prior use in other trials in similar populations.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's Disease of less than 5 years duration, with a Hoehn and Yahr stage of I-III. The diagnosis should be based on medical history and neurological examination.
2. 30 to 80 years, inclusive, at screening.
3. If female, be either post menopausal for at least 2 years, surgically sterilised or have undergone hysterectomy or, if of child bearing potential they must be willing to avoid pregnancy by using an adequate method of contraception for four weeks prior to, during and four weeks after the last dose of study medication. For the purposes of this study, women of childbearing potential are defined as all female subjects after puberty unless they are post-menopausal for at least two years, are surgically sterile or are sexually inactive.
4. Receiving treatment with a single dopamine agonist at a stable dose for at least 4 weeks prior to the screening visit.
5. Willing and able to participate in the study and have provided written, informed consent.

Exclusion Criteria:

To be eligible for inclusion in this study the subjects must not meet any of the following criteria:

1. Any indication of forms of Parkinsonism, other than idiopathic Parkinson's Disease.
2. If female, be pregnant or lactating.
3. Current diagnosis of substance abuse or history of alcohol or drug abuse in the past 3 months.
4. Currently experiencing end of dose wearing off or on-off phenomena, disabling peak dose or biphasic dyskinesias, or unpredictable or widely swinging fluctuations.
5. Current clinically significant gastrointestinal, renal, hepatic, endocrine, pulmonary or cardiovascular disease, including acute gastric ulcer, hypertension that is not well controlled, asthma, chronic obstructive pulmonary disease (COPD), and Type I diabetes. Subjects with a history of gastric ulcer who have not had a recent episode of acute gastritis and are not currently experiencing gastric pain will be eligible for inclusion.
6. Second- or third-degree atrioventricular block or sick sinus syndrome, uncontrolled atrial fibrillation, severe or unstable angina, congestive heart failure, myocardial infarction within 3 months of the screening visit, or significant ECG abnormality, including QTc ≥ 450 msec (males) or ≥ 470 msec (females), where QTc is based on Bazett's correction method.
7. Have received treatment with safinamide previously.
8. Concomitant disease likely to interfere with the study medication (e.g. capable of altering absorption, metabolism or elimination of the study drug).
9. History of, or current psychosis (e.g. schizophrenia or psychotic depression) or a score ≥ 3 on item 2 (thought disorder) or 3 (depression) of the UPDRS, Section I at screening.
10. Evidence of dementia or cognitive dysfunction, as indicated by a MMSE score < 24 or a score ≥ 3 on item 1 (mentation) of the UPDRS, Section I at screening.
11. Depression, as indicated by a GRID-HAMD (17-item scale) score > 17 at screening.
12. History of allergic response to anticonvulsants or anti-Parkinsonian agents.
13. Mental or physical condition (e.g., neurotic behaviour, crippling degenerative arthritis, or limb amputation), which would preclude performing efficacy or safety assessments.
14. Hypersensitivity or contraindications to MAO B inhibitors.
15. Current history of severe dizziness or fainting on standing, due to postural hypotension.
16. Neoplastic disorder, which is either currently active or has been in remission for less than one year.
17. Participation in a clinical trial within 30 days of entry into the trial (screening visit) or has received treatment with any investigational compound within 30 days or 5 half-lives, whichever is longer, prior to screening.
18. Treatment of their Parkinsonian symptoms with a medication, other than a stable dose of a single dopamine agonist, during the 8 weeks preceding the screening visit.
19. Treatment with any agent known to significantly inhibit or induce drug-metabolising enzymes (e.g., barbiturates, phenothiazines, etc.) within 4 weeks preceding the screening visit.
20. Treatment with opioids (e.g., tramadol, meperidine derivatives), SNRIs (e.g., venlafaxine, duloxetine), tri- or tetra-cyclic antidepressants, MAO inhibitors (e.g. selegiline), in the 8 weeks prior to the screening visit. Dextromethorphan will be permitted if used for treating cough.
21. Treatment with a depot neuroleptic within one injection cycle, or oral neuroleptics within 4 weeks prior to the screening visit.
22. Treatment with a drug that has hepatotoxic potential, e.g., tamoxifen, within 4 weeks, or received radiation therapy or a drug with cytotoxic potential, e.g., chemotherapy, within one year prior to the screening visit.
23. Diagnosis of HIV, or tests positive for Hepatitis C antibodies, or Hepatitis B surface antigen.
24. Any abnormality that the investigator deems to be clinically relevant, either on medical history, physical examination, ECG or in a diagnostic laboratory test.
25. Ophthalmologic history including any of the following conditions: albino subjects, family history of hereditary retinal disease, progressive and/or severe diminution of visual acuity (i.e., 20/70), retinitis pigmentosa, retinal pigmentation due to any cause, any active retinopathy or ocular inflammation (uveitis), or diabetic retinopathy.
26. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2007-11; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the changes from baseline to W24 in motor symptoms (UPDRS Section III). | 24 weeks

SECONDARY OUTCOMES:
Evaluate the changes from baseline to W24 in activities of daily living, cognition, change in global clinical status, responder rates with regard to motor symptoms and health related quality of life | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Willmer, MD, Study Director — Merck Serono S.A., Geneva
Locations (125):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Neurological Institute, Phoenix, Arizona
  - Pacific Neuroscience Medical Group, Oxnard, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Parkinson's Institute, Sunnyvale, California
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Parkinson's Disease and Movement Disorder Center, Boca Raton, Florida
  - Neurologic Consultants P.A., Fort Lauderdale, Florida
  - University Of Florida, Gainesville, Florida
  - Parkinson's Disease Treatment Center of SW Florida, Port Charlotte, Florida
  - Neurology Clinical Research Inc., Sunrise, Florida
  - University Of South Florida Medical Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Columbus Research Institute, Columbus, Georgia
  - Northwestern University PD and Movement Disorders Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Parkinson's Disease and Movement Disorders Center of Albany, Albany, New York
  - North Shore Medical Center, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - New York University, New York, New York
  - The Neurological Institute, Charlotte, North Carolina
  - Duke University Health Systems, Druham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Neurology Specialists, Dayton, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas
- Argentina (11):
  - Hospital Español, Buenos Aires
  - Instituto de Neurociencias Buenos Aires S.A., Buenos Aires
  - Clinica IMECO, Capital Federal
  - Hospital Italiano de Buenos Aires, Capital Federal
  - Instituto de Investigaciones Neurológicas Raul Carrea FLENI, Capital Federal
  - Instituto Frenopatico S.A., Capital Federal
  - Instituto Medico Congreso, Ciudad Autonoma de Bs. As.
  - Instituto Argentino de Investigacion Neurologica SRL, Ciudad Autonoma de
  - Instituto INEBA, Ciudad Autónoma de Bs. As.
  - Hospital Privado Centro Médico de Córdoba, Córdoba
  - Hospital Universitario Austral, Pilar
- Brazil (4):
  - Hospital das Clinicas da UFPR, Curitiba
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Centro Pediatrico Professor Hosanna de Oliveira, Salvador
  - Hospital Universitario Professor Edgard Santos - UFBA, Salvador
- Bulgaria (6):
  - CCB Medical Institute - Ministry of Interior, Sofia
  - First MHAT - Sofia AD, Sofia
  - MHAT Tokuda Hospital Sofia AD, Sofia
  - Shatcvd - Nch Ead, Sofia
  - SHATNP 'Sv. Naum' EAD, Sofia
  - UMHAT 'Tsaritsa Yoanna - ISUL' EAD, Sofia
- Canada (5):
  - Dynamik Research Inc., Pointe-Claire, Quebec
  - Kingston General Hospital, Kingston
  - Centre For Movement Disorders, Markham
  - Parkinson's and Neurodegenerative Disorders Clinic, Ottawa
  - Toronto Western Hospital - University Health Network, Toronto
- Chile (3):
  - Hospital Barros Luco Trudeau, Santiago
  - Hospital Base Valdivia, Valdivia
  - Clinica Ciudad del Mar, Viña del Mar
- Colombia (3):
  - Centro de Investigaciones del Sistema Nervioso Limitada, Bogotá
  - Fundación Clínica Abood Shaio, Bogotá
  - Instituto del Corazón, Bucaramanga
- Croatia (4):
  - Clinical Hospital Osijek, Osijek
  - Clinical Hospital Center Rijeka, Rijeka
  - Clinical Hospital "Sestre Milosrdnice", Zagreb
  - Clinical Hospital Centre Zagreb, Zagreb
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Privatni neurologicka ambulance, Hradec Králové
  - Poliklinika Modry pavilon, Ostrava
  - Clintrials.r.o., Prague
  - VFN Praha, Prague
- Finland (3):
  - Itä-Suomen yliopisto Kuopion kampus, Kuopio
  - Etelä-Karjalan keskussairaala, Lappeenranta
  - ODL Terveys Oy, Oulu
- Germany (5):
  - Charité Universitaetsmedizin Berlin - Campus Charité Mitte, Berlin
  - Ehret Reinhard, Berlin
  - St. Josef-Hospital, Berlin
  - Eberhard-Karls-Universitaet, Tübingen
  - Universitaetsklinikum Ulm, Ulm
- India (8):
  - Krishna Institute of Medical Sciences, Hyderabad
  - Nizam's Institute of Medical Sciences, Hyderabad
  - Mallikatta Neuro and Research Centre, Mangalore
  - T.N. Medical College & B.Y.L. Nair Hospital, Mumbai
  - Brain & Mind Institute, Nagpur
  - All India Institute of Medical Sciences (AIIMS), New Delhi
  - Poona Hospital & Research Center, Pune
  - Andhra Medical College, Visakhapatnam
- Italy (10):
  - AO Universitaria Policlinico di Catania, Catania
  - Fondazione Università Gabriele D'Annunzio, Chieti
  - Ospedale Versilia, Lido di Camaiore
  - Fondazione San Raffaele del Monte Tabor, Milan
  - Istituti Clinici di Perfezionamento, Milan
  - Università degli Studi "Federico II", Napoli
  - Azienda Ospedaliera Universitaria di Parma, Parma
  - IRCCS S. Raffaele Pisana, Roma
  - Ospedale San Giovanni Battista Ordine di Malta, Roma
  - Policlinico Tor Vergata, Roma
- Mexico (4):
  - Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara
  - Instituto Nacional de Neurologia, La Fama
  - Medical Sur, México
  - Instituto de Información de Investigación en Salud Mental, Monterrey
- Peru (3):
  - Hospital Alberto Sabogal Sologuren, Callao
  - Clinica Anglo Americana, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
- Pomorskie Centr.Traumatologii WSS im.M.Kopernika, Gdansk, Poland
- Hospital de Santa Maria, Lisbon, Portugal
- Slovakia (6):
  - MU Dr. Beata Dupejova Neurologicka ambulancia s.r.o, Banská Bystrica
  - FNsP Bratislava pracovisko Kramare, Bratislava
  - Poliklinika Tehelna, Bratislava
  - Vseobecna nemocnica s poliklinikou Levoca a.s., Levoča
  - Fakultna nemocnica Trnava, Trnava
  - Nestatne zdravotnicke zariadenie, Žilina
- South Africa (6):
  - Sandton Clinic, Johannesburg, Gauteng
  - Dr CC Coetzee Inc, Durban, KZ-Natal
  - Constantiaberg Medi-Clinic, Cape Town
  - Groote Schuur Hospital, Cape Town
  - St. Augustine's Medical Mews, Durban
  - Willows Medical Centre, Pretoria
- Spain (6):
  - H Clinic i Provincial, Barcelona
  - H de la Santa Creu i Sant Pau, Barcelona
  - H Mutua de Terrassa, Barcelona
  - Policlinica Guipuzcoa, Donostia / San Sebastian
  - Fundacion H. Alcorcon, Madrid
  - Fundacion Jimenez Diaz, Madrid